CLINICAL TRIAL: NCT05286541
Title: Qualitative and Quantitative Assessment of Autogenous Versus Xenogenic Horizontal Ridge Augmentation After Mandibular Ridge-split with Buccal Cortical Lateralization: a Randomizedcontrolled Trial
Brief Title: Buccal Cortical Separation and Lateralization for Horizontal Ridge Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Shawky, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OMFS 3-3-9
Record Dates: First submitted 2022-02-18; First posted 2022-03-18 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Horizontal Ridge Deficiency
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lateralized buccal cortex group with xenograft (Experimental): the buccal cortical bone was osteotomized and separated to be fixed in a lateralized position at the desired distance and the gap filled with Xenograft
  Interventions: Procedure: Lateralized buccal cortex with xenograft
- lateralized buccal cortex with autogenous particulate (Active Comparator): the buccal cortex was lateralized same as in the interventional group but the gap filled with autogenous particulate
  Interventions: Procedure: Lateralized buccal cortex with autogenous particulate

INTERVENTIONS:
Procedure: Lateralized buccal cortex with xenograft — the buccal cortex of the deficient ridge was separated and lateralized then fixed at the desired distance
  Arms: Lateralized buccal cortex group with xenograft
Procedure: Lateralized buccal cortex with autogenous particulate — lateralized buccal cortex with autogenous particulate
  Arms: lateralized buccal cortex with autogenous particulate

SUMMARY:
Cases with horizontal ridge deficiency less than what is possible for ridge splitting were recruited and the buccal cortex was totally separated and lateralized at the desired distance for augmentation

ELIGIBILITY:
Inclusion Criteria:

* suffering only from posterior mandibular horizontal ridge deficiency and with adequate inter-arch space to accommodate the future restoration

Exclusion Criteria:

* Heavy smokers, diabetics, patients with bleeding problems, liver and kidney diseases, bone diseases that can affect bone healing, previous history of any ridge augmentation procedure in the posterior mandible, and those undergoing or planned for radiotherapy or chemotherapy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Change in horizontal bone gain | six months after the operation
  the net average bone gain (in millimeters) was calculated: by calculating the difference between the immediate post operative bone width measured on the Immediate CBCT and the six months bone width measured on the six months CBCT

SECONDARY OUTCOMES:
Bone area percent | Six months after the operation
  histomorphometric analysis of core biopsies was done at the time of implant insertion to determine the bone area percent at the implant sites

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Atef, PhD, Principal Investigator — Associate Professor
Locations (1):
- Faculty of dentistry, Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Atef M, Shawky M, Mounir M, Gibaly A. Assessment of Modified Ridge Split With Autogenous Versus Xenogenic Augmentation: Randomized Clinical Trial. Clin Implant Dent Relat Res. 2025 Jun;27(3):e70046. doi: 10.1111/cid.70046. PMID 40342252